CLINICAL TRIAL: NCT03070405
Title: An Open-label, Randomized, Crossover Study to Evaluate the Effect of PAS on the Pharmacokinetics of Tenofovir in Healthy Subjects
Brief Title: The Effect of PAS on the Pharmacokinetics of Tenofovir in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Principal Investigator, Inje University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 16-0138
Record Dates: First submitted 2017-02-09; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteers
Keywords: Tenofovir Disoproxil Fumarate; 4-Aminosalicylic Acid; Tuberculosis; HIV
MeSH Terms: conditions — Tuberculosis | interventions — Tenofovir

ARMS (2):
- Tenofovir (Active Comparator): Tenofovir disoproxil fumarate 300mg single dose administration
  Interventions: Drug: Tenofovir disoproxil fumarate 300mg
- Tenofovir + PAS (Experimental): Tenofovir disoproxil fumarate 300mg single dose, Para-aminosalicylic acid Ca Granule 5.28 g BID seven dose administration
  Interventions: Drug: Tenofovir disoproxil fumarate 300mg; Drug: Para-aminosalicylic acid Ca granule 5.28 g

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate 300mg — Single oral dose on the first day of each period
  Other Names: viread
Drug: Para-aminosalicylic acid Ca granule 5.28 g — Twice daily oral administration from the first day of each period to the seventh dose
  Other Names: Pas Granule Dongindang
  Arms: Tenofovir + PAS

SUMMARY:
The main purpose of this study is to evaluate whether PAS will change the PK parameters of tenofovir.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male volunteers, ages 19 to 45 years at the time of screening test inclusive.
2. Subjects who did not have congenital or chronic diseases and sign and symptom after medical examinations
3. Body Mass Index (BMI) of 18 to 25 kg/m2, inclusive. BMI = weight (kg)/ [height (m)]2.
4. Volunteers deemed as appropriate subjects by investigators, after passing medical screening, including assessment of medical history, vital signs, 12-lead ECG, physical examination, laboratory tests etc. according to the characteristics of the investigational products.
5. Subjects who can participate in the whole clinical trial.
6. Subjects who voluntarily sign a written consent form after having received information regarding the objectives and contents of the trial, and characteristics of the study drug drugs prior to signing.

Exclusion Criteria:

1. Medical History

   1. Subjects with any disease or history of clinically significant liver, kidney, digestive system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatric system, hemato-oncologic system, urinary system, cardiovascular system including arrhythmia.
   2. Subjects with any history of gastrointestinal diseases/conditions that could impact on the absorption of study drug.
2. Laboratory Test and ECG Findings

   1. Subjects who show, or have had clinical abnormalities detected through laboratory tests prior to the trial commencement date. Criteria for liver and renal function test are shown below:

      * AST or ALT above 1.25×ULN
      * Total bilirubin above 1.5×ULN
      * Serum creatinine clearance calculated by CKD-EPI below 80mL/min
   2. Subjects who show a clinically significant abnormalities detected through ECG
3. History of hypersensitivity to the drug including study drug ingredients and other medications (aspirin, antibiotics, etc.) or clinically significant hypersensitivity
4. Prohibition on Concomitant Drug/Food

   1. Use of ethical-the-counter/herbal preparations or use of over-the-counter medications/vitamin medications within 2 weeks or 1 week prior to study drug administration, respectively
   2. Subjects on any diet which could affected study drug's pharmacokinetics
   3. Subjects who administered the Probenecid, Penicillin G and other drugs which already known has an effect on OAT1 Transporter activity within 2 weeks prior to the first dose.
5. Blood Donation and Transfusion

   1. Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 60 days prior to study drug administration.
   2. Blood transfusion within 30 days prior to study drug administration.
6. Other Exclusion Criteria

   1. Alcohol over intake (alcohol > 30g/day) and screening positive for alcohol
   2. Subjects who smoke within 3 months before initiation of clinical trial and subjects who cannot stop smoking during the participation of clinical study
   3. Subjects who cannot stop taking caffeine-containing foods (e.g. coffee, tea, green tea, cocoa, chocolate, soda, coffee milk, energy supplementary beverage, etc.) and alcoholic beverage during the participation of clinical study
   4. Subjects deemed to be inappropriate for the trial as determined by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male participants included into the study
Enrollment: 20 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of tenofovir | 0-84 hours in test and 0-72 hours in reference arm
  Cmax of Tenofovir will be compared between test and reference arms.
Area under the plasma concentration versus time curve (AUC) of tenofovir | 0-84 hours in test and 0-72 hours in reference arm
  AUC of tenofovir will be compared between test and reference arms.

SECONDARY OUTCOMES:
Volume of distribution of tenofovir | 0-84 hours in test and 0-72 hours in reference arm
Time of peak plasma concentration(Tmax) of tenofovir | 0-84 hours in test and 0-72 hours in reference arm
Plasma half-life of tenofovir | 0-84 hours in test and 0-72 hours in reference arm
Renal clearance of tenofovir | 0-24 hours
Amount of tenofovir excreted in urine | 0-24 hours
Peak plasma concentration of PAS | 0-12 hours
Area under the plasma concentration versus time curve (AUC) of PAS | 0-12 hours
Renal clearance of PAS | 0-12 hours
Volume of distribution of PAS | 0-12 hours
Time of peak plasma concentration of PAS | 0-12 hours
Plasma half-life of PAS | 0-12 hours
Amount of PAS excreted in urine | 0-12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, MD, PhD, Principal Investigator — Inje University

IPD SHARING:
Plan to Share IPD: No